CLINICAL TRIAL: NCT03742765
Title: Incentivizing Planning & Output in Exercising
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 827107-1255
Record Dates: First submitted 2018-11-13; First posted 2018-11-15 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Healthy
Keywords: Exercise; Incentives; Planning
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incentivizing Planning (Experimental): Participants will receive three texts each week asking a question to help plan for the next workout, and will receive 500 points for each text they answer. These bonus points are on top of points participants receive for each workout (200 points per workout).
  Interventions: Behavioral: Incentivizing planning
- Incentivizing Exercise (Experimental): Participants will receive three texts each week asking a question about their workout. Regardless of whether or not they respond to the texts, participants receive 500 bonus points for their first three workouts during the week. These bonus points are on top of points participants receive for each workout (200 points per workout).
  Interventions: Behavioral: Incentivizing exercise

INTERVENTIONS:
Behavioral: Incentivizing planning — Participants receive bonus incentives for planning their workouts
  Arms: Incentivizing Planning
Behavioral: Incentivizing exercise — Participants receive bonus incentives for exercising
  Arms: Incentivizing Exercise

SUMMARY:
This study will test whether incentivizing pre-workout activities (i.e., planning workouts) is more effective than incentivizing actual workouts. This study has two conditions: planning condition (with incentives for planning) vs. output (with incentives for working out). The focus of the incentives will be reinforced by three text messages per week and weekly emails.

DETAILED DESCRIPTION:
Gym members register online to participate in a 28-day workout program. Upon registration, participants are assigned to one of two conditions (a condition that incentivizes planning or a condition that incentivizes workouts). Upon registration, participants are prompted to create a workout schedule and are given tips about how to create a workout habit. Over the 28-day intervention period, participants receive text message reminders prior to their scheduled workouts and emails reminding them of their schedules. In both conditions, participants receive points every day that they go to the gym, which can be redeemed for a gift card after the intervention period. In the planning condition, participants can receive bonus points for responding to each of three text messages each week asking about their plans for going to the gym. In the output condition, participants receive bonus points for their first three workouts each week.

ELIGIBILITY:
Inclusion Criteria:

* Has 24 Hour Fitness gym membership

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Gym visits per week | During the 28-day intervention period
  Number of times the participant goes to the gym
Gym visits per week | During the 4-weeks post-intervention
  Number of times the participant goes to the gym
Gym visits per week | During the 10-weeks post-intervention
  Number of times the participant goes to the gym
Whether or not a participant visits the gym in a given week | During the 28-day intervention period
  Binary variable capturing whether or not a participant had any gym visits in a given week
Whether or not a participant visits the gym in a given week | During the 4-weeks post intervention
  Binary variable capturing whether or not a participant had any gym visits in a given week
Whether or not a participant visits the gym in a given week | During the 10-weeks post intervention
  Binary variable capturing whether or not a participant had any gym visits in a given week

SECONDARY OUTCOMES:
Gym visits per week | During the 52-weeks post-intervention
  Number of times the participant goes to the gym
Whether or not a participant visits the gym in a given week | During the 52-weeks post-intervention
  Binary variable capturing whether or not a participant had any gym visits in a given week

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No